CLINICAL TRIAL: NCT02898428
Title: Continuous Glucose Monitoring During Breastfeeding or Formula Feeding in New Mothers With Type 1 Diabetes
Brief Title: Continuous Glucose Monitoring in New Mothers With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Principal Investigator, Lene Ringholm, Chief physician, Steno Diabetes Center Copenhagen
Other Study IDs: SDC-2016-055
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Hypoglycemia; Breastfeeding
MeSH Terms: conditions — Hypoglycemia; Breast Feeding | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- New mothers: New mothers with type 1 diabetes
  Interventions: Device: Continuous glucose monitoring (CGM)
- Control group: Non-pregnant, non-breastfeeding women with type 1 diabetes matched for age and BMI
  Interventions: Device: Continuous glucose monitoring (CGM)

INTERVENTIONS:
Device: Continuous glucose monitoring (CGM)

SUMMARY:
With appropriate day-time carbohydrate intake and insulin dose, the 24 hour glucose levels and prevalence of night-time hypoglycaemia are comparable in breastfeeding new mothers and formula feeding new mothers with type 1 diabetes at the second after delivery diabetes control compared with the first after delivery diabetes control at Steno Diabetes Center.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years.
* Delivery of a single infant.
* Proficiency in Danish to read and understand the patient information sheet, questionnaires and to converse with the diabetes caregivers.

Exclusion Criteria:

* A diagnosis with severe mental or psychiatric barriers or a concurrent disease on the decision of the principal investigator

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: New mothers with type 1 diabetes
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Hypoglycemia | Night-time 8 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Denmark

REFERENCES:
- [Derived] Ringholm L, Roskjaer AB, Engberg S, Andersen HU, Secher AL, Damm P, Mathiesen ER. Breastfeeding at night is rarely followed by hypoglycaemia in women with type 1 diabetes using carbohydrate counting and flexible insulin therapy. Diabetologia. 2019 Mar;62(3):387-398. doi: 10.1007/s00125-018-4794-9. Epub 2019 Jan 3. PMID 30607466